CLINICAL TRIAL: NCT01152892
Title: Risk Stratification in End Stage Renal Disease (ISAR)
Brief Title: Risk Stratification in End Stage Renal Disease (ESRD) - ISAR Study
Acronym: ISAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Else Kröner Fresenius Foundation (Other); AIT Austrian Institute of Technology GmbH (Other); Ludwig-Maximilians - University of Munich (Other); FH Aachen, University of applied sciences (Unknown)
Responsible Party: Principal Investigator, PD Dr. Christoph Schmaderer, PD Dr. med. Christoph Schmaderer, Technical University of Munich
Other Study IDs: ISAR ESRD 01 2010
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: End Stage Renal Disease; Chronic Kidney Disease; Cardiovascular Event; Sudden Cardiac Death
Keywords: end stage renal disease; chronic kidney disease; cardiovascular event; sudden cardiac death; autonomic function
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the use of non-invasive markers of the autonomic function and micro- and macrocirculation to predict mortality and cardiovascular end points in end-stage renal disease patients. Furthermore we aim at getting new insight into the insufficiently understood pathophysiology leading to excessively high cardiovascular and non-cardiovascular mortality in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. End-stage renal disease (ESRD) and receiving maintenance hemodialysis

Exclusion Criteria:

1. Any clinically significant infection.
2. pregnancy
3. history of malignant disease with a prognostic life expectancy less than 24 months
4. missing of written and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with end stage renal disease treated with chronic hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-04; Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Mortality of all causes | 24 months
  24 month follow up

SECONDARY OUTCOMES:
Incidence of cardiovascular events | 24 months
  24 month follow up
Blood pressure drops within a dialysis session | 24 months
  24 month follow up
Incidence of infections requiring antibiotic treatment | 24 months
  24 month follow up
Incidence of shunt thrombosis | 24 months
  24 month follow up
incidence of death and hospitalization due to infection | 24 months
  24 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schmaderer, M.D., PD, Principal Investigator — study chief investigator and head of the nephrological laboratory at the department of nephrology of the Klinikum rechts der Isar of the Technical University of Munich
Locations (17):
- Germany (17):
  - KFH Dialysis Center, Altötting, Bavaria
  - KFH Dialysis Center Dillingen, Dillingen an der Donau, Bavaria
  - Praxen Dr. Braun Dingolfing, Dingolfing, Bavaria
  - KFH Dialysis Center Elsenheimerstrasse, Munich, Bavaria
  - KFH Dialysis Center Munich Schwabing, Munich, Bavaria
  - KFH Dialysis Center Munich Harlaching, Munich, Bavaria
  - KFH Dialysis Center Neuried, Munich, Bavaria
  - Dialysezentrum München Nord, München, Bavaria
  - Dialysezentrum München Solln, München, Bavaria
  - KFH Nierenzentrum Giesinger Bahnhof, München, Bavaria
  - Department of nephrology, Klinikum rechts der Isar, München, Bavaria
  - Nierenzentrum Perlach, München, Bavaria
  - Nierenzentrum Bogenhausen, München, Bavaria
  - KFH Dialysis Center Oberschleißheim, Oberschleißheim, Bavaria
  - KFH Dialysis Center Unterhaching, Unterhaching, Bavaria
  - KFH Dialysis Center Weißenburg, Weißenburg in Bayern, Bavaria
  - Dialyse im Zentrum, München

REFERENCES:
- [Background] Bauer A, Kantelhardt JW, Barthel P, Schneider R, Makikallio T, Ulm K, Hnatkova K, Schomig A, Huikuri H, Bunde A, Malik M, Schmidt G. Deceleration capacity of heart rate as a predictor of mortality after myocardial infarction: cohort study. Lancet. 2006 May 20;367(9523):1674-81. doi: 10.1016/S0140-6736(06)68735-7. PMID 16714188
- [Derived] Werfel S, Gunthner R, Hapfelmeier A, Hanssen H, Kotliar K, Heemann U, Schmaderer C. Identification of cardiovascular high-risk groups from dynamic retinal vessel signals using untargeted machine learning. Cardiovasc Res. 2022 Jan 29;118(2):612-621. doi: 10.1093/cvr/cvab040. PMID 33576412
- [Derived] Gunthner R, Hanssen H, Hauser C, Angermann S, Lorenz G, Kemmner S, Matschkal J, Braunisch MC, Kuechle C, Renders L, Moog P, Wassertheurer S, Baumann M, Hammes HP, Mayer CC, Haller B, Stryeck S, Madl T, Carbajo-Lozoya J, Heemann U, Kotliar K, Schmaderer C. Impaired Retinal Vessel Dilation Predicts Mortality in End-Stage Renal Disease. Circ Res. 2019 Apr 1. doi: 10.1161/CIRCRESAHA.118.314318. Online ahead of print. PMID 30929571
- [Derived] Hagmair S, Braunisch MC, Bachler M, Schmaderer C, Hasenau AL, Bauer A, Rizas KD, Wassertheurer S, Mayer CC. Implementation and verification of an enhanced algorithm for the automatic computation of RR-interval series derived from 24 h 12-lead ECGs. Physiol Meas. 2017 Jan;38(1):1-14. doi: 10.1088/1361-6579/38/1/1. Epub 2016 Dec 12. PMID 27941217
- [Derived] Schmaderer C, Tholen S, Hasenau AL, Hauser C, Suttmann Y, Wassertheurer S, Mayer CC, Bauer A, Rizas KD, Kemmner S, Kotliar K, Haller B, Mann J, Renders L, Heemann U, Baumann M. Rationale and study design of the prospective, longitudinal, observational cohort study "rISk strAtification in end-stage renal disease" (ISAR) study. BMC Nephrol. 2016 Oct 26;17(1):161. doi: 10.1186/s12882-016-0374-8. PMID 27784272